CLINICAL TRIAL: NCT02608060
Title: Open Multicentric Study to Assess the Hematopoyetic Response in Terms of Increase of Hemoglobin Levels of Patients With Anemia Related to Non- Hodgkin Lymphoma, Chronic Lymphocytic Leukemia or Multiple Myeloma, Treated With Erythropoietin B (Recormon) Using Pre-filled Syringe With 30000 IU, as Well as to Quantify the Risk Factors of Anemia and Its Impact on Quality of Life Related to Treatment
Brief Title: A Study to Assess the Hematopoyetic Response of Anemic Patients With Hematologic Malignancies Treated With Erythropoietin B
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to poor enrollment this study was terminated prematurely.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18055
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta

ARMS (1):
- Epoetin Beta - 30000 IU (Experimental): Dosage at Initiation: Subcutaneous injection of 30000 IU epoetin beta administered once a week. Dosage could be increased to 30000 IU twice a week or 60000 IU once a week after 4 weeks if a blood transfusion was required or hemoglobin level did not increase by at least 0.5 grams per deciliter (g/dL) versus baseline.
  Interventions: Drug: Epoetin Beta

INTERVENTIONS:
Drug: Epoetin Beta — Dosage at Initiation: Subcutaneous injection of 30000 IU administered once a week. Dosage could be increased to 30000 IU twice a week or 60000 IU once a week after 4 weeks if a blood transfusion was required or hemoglobin level did not increase by at least 0.5 g/dL versus baseline.
  Other Names: Recormon

SUMMARY:
This study will examine the efficacy, safety and effect on hemoglobin levels, of once weekly subcutaneous injections of epoetin beta (30,000 IU) in anemic participants with non-Hodgkin's lymphoma, chronic lymphocytic leukemia or multiple myeloma. The anticipated study duration is 4 months, and the target sample size is 30 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with a diagnosis of non-Hodgkin's lymphoma, chronic lymphocytic leukemia or multiple myeloma
* Anemia at Screening Visit

Exclusion Criteria:

* Transfusion of red blood cells within 2 months of study drug
* Treatment-resistant hypertension
* Acute or chronic bleeding (requiring therapy) within 3 months of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Hemoglobin levels at 16 weeks | 16 Weeks

SECONDARY OUTCOMES:
Serum Iron, Ferritin and Transferrin Levels | 16 Weeks
Time to Global Response | Up to 4 months
Percentage of Participants with a Positive Response | Weeks 4 and 8
Quality of Life in Relation to Grade of Anemia | Up to 4 months
Quality of Life According to the Functional Assessment of Cancer Therapy - Anemia (FACT-An) Instrument | Up to 4 months
Tolerability - Incidence of Adverse Events | Up to 16 Weeks of treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Caracas, Venezuela